CLINICAL TRIAL: NCT05716256
Title: Effect of Ulinastatin on the Action of Nondepolarising Muscle Relaxants Rocuronium / Cisatracurium
Brief Title: Effect of Ulinastatin on the Action of NDMRs (Rocuronium / Cisatracurium)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ai Ling, Ai Ling, Doctor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TJ-IRB20221241
Record Dates: First submitted 2023-01-12; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Nondepolarising Muscle Relaxants
Keywords: Ulinastatin; Rocuronium; Cisatracurium; Train of four (TOF)
MeSH Terms: interventions — urinastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulinastatin (Experimental): The experimental groups （Rocuronium-Ulinastatin group and Cisatracurium-Ulinastatin group）received ulinastatin 5000U/kg followed by rocuronium 0.6 mg/kg or cisatracurium 0.1 mg/kg
  Interventions: Drug: Ulinastatin; Procedure: TOF monitoring
- Conventional treatment group (Sham Comparator): The control groups（Rocuronium-Saline group and Cisatracurium-Saline group） received normal saline 0.1ml/kg followed by rocuronium 0.6 mg/kg or cisatracurium 0.1 mg/kg
  Interventions: Drug: Ulinastatin; Procedure: TOF monitoring

INTERVENTIONS:
Drug: Ulinastatin — The CIS-ULI group received ulinastatin 5000U/kg followed by cisatracurium 0.1 mg/kg The CIS-NS (control) group received normal saline 0.1ml/kg followed by cisatracurium 0.1 mg/kg. The ROC-ULI group received ulinastatin 5000U/kg followed by rocuronium 0.6 mg/kg The ROC-NS (control) group received normal saline 0.1ml/kg followed by rocuronium 0.6 mg/kg
Procedure: TOF monitoring — The acceleromyograph TOF-Watch® SX (Organon, Ireland) is used for TOF monitoring. When the Narcotrend™ index is below 50 and level of anesthesia assessed as deep enough, TOF stimulation is started at 50 mA amplitudes and the setup is checked for any problem concerning the electrodes impedance and local hand temperature. After 1 minute, TOF stimulation is stopped and a tetanic stimulation (each electrical stimulus of 200μs duration and 50 mA amplitude) is delivered at a frequency of 50Hz for 5 seconds. After this procedure the alignment of sensors are checked to see if they are intact and readjust to their initial position if necessary. A no stimulation pause is observed during 3 minutes.

SUMMARY:
The aim of this research was to determine the influence of ulinastatin on nondepolarising muscle relaxants Rocuronium and Cisatracurium.

DETAILED DESCRIPTION:
BACKGROUND: Ulinastatin is a protease inhibitor derived from human urine. The effects of ulinastatin on muscle relaxants have been attributed to its capacities to cause increase in liver circulation, diuresis and possibly increased acetylcholine release. Rocuronium is mainly eliminated via the liver and kidneys whereas cisatracurium is mainly cleared via Hofmann elimination which is organ independent. The effects of ulinastatin on cisatracurium have not been assessed before. Moreover the effects of ulinastatin on the recovery period of rocuronium have not been adequately studied before. In this study, the effects of ulinastatin on cisatracurium are compared with the effects of ulinastatin on rocuronium. This is done by contrasting the ulinastatin induced changes in onset time, clinical duration and recovery duration for rocuronium with those for cisatracurium.

METHODS: 80 patients will be enrolled in this study and assigned randomly into 4 equal groups. The ROC-ULI group received ulinastatin 5000U/kg followed by rocuronium 0.6 mg/kg, the ROC-NS (control) group received normal saline 0.1ml/kg followed by rocuronium 0.6 mg/kg, the CIS-ULI group received ulinastatin 5000U/kg followed by cisatracurium 0.1 mg/kg and the CIS-NS (control) group received normal saline 0.1ml/kg followed by cisatracurium 0.1 mg/kg. The time lag between either ulinastatin or normal saline administration and muscle relaxant injection is 2 minutes. Acceleromyography using response to TOF (train of four) stimulation is used to assess neuromuscular function. The site of stimulation and response assessment are the ulnar nerve and the adductor pollicis muscle respectively. The time parameters assessed in each group are the onset time, the times to return of the first, second, third and fourth response to TOF stimulation (RT1, RT2, RT3 and RT4 respectively), the duration of moderate neuromuscular block (RT1-RT4), the duration 25% (clinical duration), the duration 50%, the recovery TOF 0.7 period and the duration TOF 0.7. Anesthesia is induced and maintained with propofol using target controlled infusion. Analgesia is achieved with an initial bolus of sufentanil followed by remifentanil infusion. Depth of anesthesia is monitored using the Narcotrend™ index. p < 0.05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo elective pancreaticoduodenectomy surgery
2. Age ranging from 25 to 60 years，body mass index (BMI)18-24kg/m2, American Society of Anesthesiologists (ASA) grades 1 or 2.
3. Receive general anesthesia and muscle relaxants intraoperatively.

Exclusion Criteria:

1. patients ASA class 3 and above
2. Severe cardiac or respiratory diseases, liver or kidney disease
3. Pregnant women.
4. Patients with neurological dysfunction including myasthenia gravis, epilepsy or psychiatric disorders
5. Patients on any premedications including antisialagogues .
6. Patients on drugs known to interfere with neuromuscular transmission including but not exclusive to anticonvulsants, calcium channel blockers, β-blockers, corticosteroids, diuretics and antibiotics of the aminoglycoside group
7. Patients known allergy to propofol and sufentanil or remifentanil,
8. emergency operations.
9. Patients judged by the investigator to be unsuitable for participation in this study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Onset time | 1 day
  Onset time defined as the period from start of injection of neuromuscular blocker to the time point when T1 has depressed to 5% of its initial control value.
RT1 | 1 day
  RT1 defined as the time from start of injection of neuromuscular blocker to T1 reappearance.
RT2 | 1 day
  Duration of moderate neuromuscular block (RT1-RT4)
RT3 | 1 day
  RT3 defined as the time from start of injection of neuromuscular blocker to T3 reappearance
RT4 | 1 day
  RT4 defined as the time from start of injection of neuromuscular blocker to T4 reappearance
Duration of moderate neuromuscular block (RT1-RT4) | 1 day
  Duration of moderate neuromuscular block (RT1-RT4) defined as the time from reappearance of T1 to reappearance of T4.
Duration 25% | 1 day
  Duration 25% defined as the time from start of injection of neuromuscular blocker to T1 recovery to 25%.
Duration 50% | 1 day
  Duration 50% defined as the time from start of injection of neuromuscular blocker to T1 recovery to 50%.
Duration TOF 0.7 | 1 day
  Duration TOF 0.7 defined as the time from start of neuromuscular blocker injection to recovery of TOF ratio to 0.7.
Recovery TOF 0.7 period | 1 day
  Recovery TOF 0.7 period defined as the time from reappearance of T4 to recovery of TOF ratio to 0.7.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Hui, Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China